## Interindividual Postexercise Hypotension Response in Morbid

NCT05504629

**Obesity** 

Date: March 17th, 2021

## **Study documents**

**Scientific background:** Physical inactivity and sedentary behaviour [i.e., Do not adhere to international physical activity guidelines of a minimum of 150 min of physical activity <sup>1</sup>] together with other lifestyle conditions (i.e., unhealthy nutrition, or poor sleep time) promote obesity, and cardiometabolic diseases such as type to diabetes mellitus (T2DM), and arterial hypertension (HTN) 2, two major diseases in the modernity, and of high prevalence in populations with excessive of adiposity such as those with morbid obesity <sup>2</sup>. Unfortunately, metabolic syndrome (MetS), another more complex cardiometabolic square that implies also obesity, poor glucose control, high blood pressure, dyslipidaemia, and high triglycerides in plasma exacerbates the risk for suffering from cardiovascular disease particularly those with morbid obesity who are candidates for bariatric surgery<sup>3</sup>. For example, a relevant meta-analysis of 87 studies with a sample of (n=951.083) showed that MetS risk factors were associated with an increased risk for cardiovascular disease (CVD) (Relative Risk, [RR]= 2.35), CVD mortality (RR= 2.40), myocardial infarction (RR= 1.99, stroke (RR= 2.27), and all-cause mortality (RR= 1.58) 4. Patients with Morbid obesity are a particular population that suffers from multiple risks for CVD, including MetS, endothelial dysfunction, as well as HTN and T2DM risk factors, all of these related to a better or worse profile to deal with success and better recovery period after bariatric surgery <sup>1</sup>. From the National Health Survey of Chile, there was described that morbid obesity is a worrying concern in women in childbearing ages 20 to 45 y, showing almost no changes from 2003 (2.2%) to 2009-10 Survey (2.1%) <sup>5</sup>. Thus, among these patients, to acquire the bariatric surgery benefit, these increase their possibilities to lose excess weight near to ~50%, to recover their overall cardiometabolic health <sup>6</sup>, and this has been strongly related to improvements in their quality o life <sup>7</sup>.

From here, lifestyle interventions such as exercise training play a key role 8-10, and relevant international organizations such as the American College of Sports Medicine <sup>1</sup>, and the European Association For The Study of Obesity Physical Activity Working Group <sup>11</sup> have recently highlighted their benefits before and after bariatric surgery. Exercise training is a known but poorly used strategy for controlling cardiometabolic risk in populations with T2DM, HTN, and MetS 8,12. At least in the blood pressure, and vascular context, exercise training decrease chronic, and acute blood pressure levels <sup>13-16</sup>. For example, a single session of endurance training (ET) (also known as moderateintensity continuous training), decreased the 24 h blood pressure <sup>17</sup>, being the magnitude of this effect is superior in subjects with higher blood pressure (systolic [SBP]/diastolic [DBP] –16.1/–7.5 mmHg) <sup>17</sup> and to those with HTN controlled and HTN not so controlled <sup>18,19</sup>, but clearly, less marked in healthy normotensive subjects (SBP/DBP -5.6/-3.1 mmHg) <sup>20</sup>. These effects have been confirmed by relevant meta-analysis where long-term ET has been a recognized strategy to get these goals in pre- and hypertensive populations <sup>21,22</sup>. On the other hand, RT also decreases blood pressure, where only 45 minutes after an acute resistance training (RT) session in HTN subjects (SBP/DBP -22.0/-8.0 mmHg), and this have been also confirmed by other relevant meta-analyses where summarize blood pressure decreases after RT in -4.4 mmHg <sup>23</sup>. Recently, and in similar coherence with ET, the RT modality has reported higher magnitude in BP reduction in subjects with elevated (SBP/DBP -12.0/-4.0 mmHg), than healthy subjects (SBP/DBP -4.0/-1.0 mmHg) <sup>24</sup>. From here, the postexercise hypotension (PEH) [i.e., defined as a reduction in systolic and/or diastolic arterial blood below control levels after a single but of exercise <sup>25</sup>] is the first vascular benefits immediately after exercise adquire a meaningful relevance, in terms that the summary of physiological adaptations by each exercise session can promote a renoval of the vasculature structure using molecular mechanisms <sup>26</sup>. Thus, as after both ET and RT, there are a number of evidence reporting the PEH benefits in different cohorts, but unfortunately there is little evidence reporting this phenomenon after concurrent training (CT), and yet less knowledge in population with MetS risk factors, as those with morbid obesity.

On the other hand, the main PEH studies report data in terms of 'average data', and it is well known that there is a wide interindividual variability to exercise training <sup>27</sup>, being a need for the report of data at an individual level. Thus, considering that there is little knowledge about the role of the order (i.e., starting by ET plus RT or by RT plus ET) in the CT session, taking into account that risk factors for MetS increase the risk for vascular damage and CVD. This study will follow the CONSORT guidelines for randomised trials, will be developed in accordance with the Declaration of Helsinki (2013), and has been approved by the Ethical Committee of the Universidad de La Frontera, Temuco, Chile (DI18-0043 Project, ACTA Nº 080 21). Design: A quasiexperimental clinical study. Methods: Patients with morbid obesity were invited for participating by a public invitation and directly to the Morbidly Obesity Association of Temuco, City, Chile (OBEMOB). After providing wide information and feedback about the risks/benefits of the intervention, all participants signed informed consent for participating in the study. We recruited diagnosed morbid obesity sedentary/physically inactive subjects (body mass index [BMI] between ≥40 kg/m<sup>2</sup>; aged 30 to 55 years) that were under the OBEMOB institution, who were assigned for convenience in 1:1 allocation to a CT group of endurance [ET] plus resistance training [RT] (ET+RT; n=17; BMI 47.8 $\pm$ 16.7) or resistance training plus endurance training group (RT+ET; n=13; BMI 43.0±8.0). Patients were recruited between 2020 and 2021 year from the above nongovernmental mentioned institution. All participants were part of the lifestyle program

previous to the possibility of receiving the bariatric surgery benefit for this disease condition from the Health Ministry of Chile (MINSAL).

## REFERENCES

- 1. Kanaley JA, Colberg SR, Corcoran MH, et al. Exercise/Physical Activity in Individuals with Type 2 Diabetes: A Consensus Statement from the American College of Sports Medicine. *Medicine and science in sports and exercise* 2022; **54**(2): 353-68.
- 2. Booth FW, Roberts CK, Laye MJ. Lack of exercise is a major cause of chronic diseases. *Comprehensive Physiology* 2012; **2**(2): 1143-211.
- 3. Bellicha A, van Baak MA, Battista F, et al. Effect of exercise training before and after bariatric surgery: A systematic review and meta-analysis. *Obesity Reviews* 2021; **22**: e13296.
- 4. Mottillo S, Filion KB, Genest J, et al. The metabolic syndrome and cardiovascular risk: a systematic review and meta-analysis. *Journal of the American College of Cardiology* 2010; **56**(14): 1113-32.
- 5. Araya M, Padilla O, Garmendia ML, Atalah E, Uauy R. Obesidad en mujeres chilenas en edad fértil. *Revista médica de Chile* 2014; **142**(11): 1440-8.
- 6. Deitel M, Shahi B. Morbid obesity: selection of patients for surgery. *Journal of the American College of Nutrition* 1992; **11**(4): 457-62.
- 7. Sierżantowicz R, Ładny JR, Lewko J. Quality of Life after Bariatric Surgery—A Systematic Review. *International Journal of Environmental Research and Public Health* 2022; **19**(15): 9078.
- 8. Flück M. Functional, structural and molecular plasticity of mammalian skeletal muscle in response to exercise stimuli. *Journal of Experimental Biology* 2006; **209**(12): 2239-48.

- 9. Delgado-Floody P, Izquierdo M, Ramírez-Vélez R, et al. Effect of High-Intensity Interval Training on Body Composition, Cardiorespiratory Fitness, Blood Pressure, and Substrate Utilization During Exercise Among Prehypertensive and Hypertensive Patients With Excessive Adiposity. *Frontiers in Physiology* 2020; **11**.
- 10. Floody PD, Lizama AC, Hormazábal MA, Poblete AO, Navarrete FC, Mayorga DJ. Evaluation of a comprehensive program of four months of duration on the preoperative conditions of obese patients candidates for bariatric surgery. *Nutricion hospitalaria* 2015; **32**(3): 1022-7.
- 11. Oppert JM, Bellicha A, van Baak MA, et al. Exercise training in the management of overweight and obesity in adults: Synthesis of the evidence and recommendations from the European Association for the Study of Obesity Physical Activity Working Group. *Obesity Reviews* 2021; **22**: e13273.
- 12. Booth FW, Chakravarthy MV, Gordon SE, Spangenburg EE. Waging war on physical inactivity: using modern molecular ammunition against an ancient enemy. *Journal of Applied Physiology* 2002; **93**(1): 3-30.
- 13. Bonsu B, Terblanche E. The training and detraining effect of high-intensity interval training on post-exercise hypotension in young overweight/obese women. *European journal of applied physiology* 2016; **116**(1): 77-84.
- 14. Álvarez C, Olivo, J., Robinson, O., Quintero, J., Carrasco, V., Ramírez-Campillo, R., Andrade, D.C., y Martínez, C. Respuesta hipotensiva de la presión sistólica y diastólica a una sesión de ejercicio aeróbico en niños, adolescentes y adultos. *Revista Medica de Chile* 2013; **141**.
- 15. Cano-Montoya J, Mancilla-Ramirez K, Cenzano L, et al. EFECTO AGUDO DE EJERCICIO ISOMÉTRICO SOBRE LA PRESIÓN ARTERIAL EN ADOLESCENTES

- CON SOBREPESO Y OBESIDAD. *Journal of Sport and Health Research* 2021; **13**(Supl 1): 51-64.
- 16. Cornelissen VA, Fagard RH. Effects of endurance training on blood pressure, blood pressure–regulating mechanisms, and cardiovascular risk factors. *Hypertension* 2005; **46**(4): 667-75.
- 17. Karoline de Morais P, Sales MM, Alves de Almeida J, Motta-Santos D, Victor de Sousa C, Simões HG. Effects of aerobic exercise intensity on 24-h ambulatory blood pressure in individuals with type 2 diabetes and prehypertension. *Journal of Physical Therapy Science* 2015; **27**(1): 51-6.
- 18. Ciolac EG, Guimarães GV, Bortolotto LA, Doria EL, Bocchi EA. Acute aerobic exercise reduces 24-h ambulatory blood pressure levels in long-term-treated hypertensive patients. *Clinics* 2008; **63**(6): 753-8.
- 19. Ciolac EG, Guimarães GV, Bortolotto LA, Doria EL, Bocchi EA. Acute effects of continuous and interval aerobic exercise on 24-h ambulatory blood pressure in long-term treated hypertensive patients. *International journal of cardiology* 2009; **133**(3): 381-7.
- 20. Park S, Rink LD, Wallace JP. Accumulation of physical activity leads to a greater blood pressure reduction than a single continuous session, in prehypertension. *Journal of Hypertension* 2006; **24**(9): 1761-70 10.097/01.hjh.0000242400.37967.54.
- 21. Montero D, Roche E, Martinez-Rodriguez A. The impact of aerobic exercise training on arterial stiffness in pre-and hypertensive subjects: a systematic review and meta-analysis. *International journal of cardiology* 2014; **173**(3): 361-8.
- 22. Cornelissen VA, Smart NA. Exercise training for blood pressure: a systematic review and meta-analysis. *J Am Heart Assoc* 2013; **2**(1): e004473.

- 23. Kelley GA, Kelley KS. Progressive Resistance Exercise and Resting Blood Pressure: A Meta-Analysis of Randomized Controlled Trials. *Hypertension* 2000; **35**(3): 838-43.
- 24. Farinatti P, Polito MD, Massaferri R, et al. Postexercise hypotension due to resistance exercise is not mediated by autonomic control: A systematic review and meta-analysis. *Autonomic Neuroscience* 2021; **234**: 102825.
- 25. Kenney MJ, Seals DR. Postexercise hypotension. Key features, mechanisms, and clinical significance. *Hypertension* 1993; **22**(5): 653-64.
- 26. La Favor JD, Dubis GS, Yan H, et al. Microvascular endothelial dysfunction in sedentary, obese humans is mediated by NADPH oxidase: influence of exercise training. *Arteriosclerosis, thrombosis, and vascular biology* 2016; **36**(12): 2412-20.
- 27. Bouchard C, Rankinen T. Individual differences in response to regular physical activity. *Medicine and science in sports and exercise* 2001; **33**(6 Suppl): S446-51.
- 28. Hopkins WG, Marshall SW, Batterham AM, Hanin J. Progressive statistics for studies in sports medicine and exercise science. *Medicine and science in sports and exercise* 2009; **41**(1): 3-13.
- 29. Green DJ, Eijsvogels T, Bouts YM, et al. Exercise training and artery function in humans: nonresponse and its relationship to cardiovascular risk factors. *Journal of Applied Physiology* 2014; **117**(4): 345-52.

**Statistical Analysis Plan (SAP):** Data are presented as the mean ± standard deviation (SD). Normality and homoscedasticity assumptions for all data were checked using the Shapiro-Wilk and Levene tests. Wilcoxon's test was used for non-parametric data. After this, we performed 2-way ANOVA (group x time) to test SBP, DBP, MAP, HR, and PP outcomes in absolute values, where Sidac's *post hoc* was applied to identify

potential differences between ET+RT vs. RT+ET. Additionally, delta changes (Δ) from pre-post were calculated to SBP, DBP, MAP, HR, and PP outcomes to test by the independent Student t-test differences between groups, where optionally the nonparametric Wilcoxon test was applied for non-parametric variables. The Cohen d effect size was obtained with threshold values at 0.20, 0.60, 1.2, and 2.0 for small, moderate, large, and very large effects, respectively <sup>28</sup>. These analyses were carried out by the statistical software Graph Pad Prism 8.0 software (Graph Pad Software, San Diego, CA, USA). After this, all results in  $\Delta$  changes of the sum of SBP  $\Sigma \Delta$ SBP was individualized and presented in quartile to be categorized in those participants 'nonresponders' (NRs; Q1 with SBP < -1 mmHg), 'low' responders (LRs; Q2 with SBP -1 to -9.9 mmHg), 'moderate' responders (MRs; Q3 with SBP -10 to -18 mmHg), and 'high' responders (HRs; Q4 with SBP  $\geq -18$  mmHg) according with their blood pressure changes (i.e., particularly decreases) as previously have been reported <sup>29</sup>. Linear regression was applied in the backward mode for testing those potential body composition, metabolic and physical condition outcomes predictors outcomes of the PEH. The  $\sum \Delta SBP$  decreases an average of the session 1 and 2 of both ET+RT and RT+ET groups related to the PEH (i.e., decreases in SBP) was used as 'dependent' outcome, while age, height, body mass, BMI, waist circumference, body fat in % and kg, lean mass, skeletal muscle mass, bone mass, total body water, BMR, SBP, DBP, HR at rest, pulse pressure, fasting glucose, total cholesterol, LDL-c, HDL-c cholestetrol, triglycerides, 6Mwt, and handgrip muscle strength (dominan, and non-dominant arm) were used as 'independent' predictors. Statistical analyses for these procedures were applied using SPSS software version 28 (SPSS<sup>TM</sup> Inc., Chicago, Illinois, USA). The alpha level was fixed at (p<0.05) for all tests of statistical significance.